CLINICAL TRIAL: NCT02553993
Title: Comparing the Cognitive Effects of Two Exergame Balance Training Systems and Traditional Weight Shifting Training in Patients With Chronic Stroke
Brief Title: Comparing the Cognitive Effects of Two Exergame Training and Traditional Training in Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG8C0261
Record Dates: First submitted 2015-09-14; First posted 2015-09-18 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-09

CONDITIONS: Stroke
Keywords: Stroke; Cognition; Exergames; Weight shifting; Balance; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Wii Fit (Experimental): The Wii Fit training was conducted using the Wii Fit bundle from Nintendo, which consists of the Wii console, a Wii Balance Board, and the Wii Fit Plus balance game disc. The Wii balance board has 4 transducers, which could assess the player's force distribution and resultant movements in the center of pressure (COP). The participants stood on the board and used the change of COP to play the games. Five games (Tilt, Soccer Heading, Balance Bubble, Penguin Slide, and Perfect 10) were selected from the Wii Fit Plus package based on the motor demand of these games. The major movement patterns to play the games included right-left weight shifting and front-back weight shifting.
  Interventions: Device: Wii Fit(30 Mins)
- Tetrax biofeedback (Experimental): The Tetrax biofeedback games aimed at postural rehabilitation to help patients or athletes improve their balance abilities. There were 11 games in Tetrax system; 8 games (Speedtrack, Catch, Skyball, Gotcha, Speedball, Tag, Freeze, Immobilizer) were chosen based on the same principle as those used for choosing Wii Fit games. The parameters of games' difficulties included target size and/or speed of target movement, which could be adjusted according to the patients' ability.
  For the Wii Fit or Tetrax group, at each session, the supervising therapist chose 3 to 5 games for participants according to their ability, needs, and favorites.
  Interventions: Device: Tetrax biofeedback(30 Mins)
- Conventional weight-shifting (Placebo Comparator): The conventional weight-shifting exercise group performed balance exercises with the similar movements and time required by the 2 exergame systems but without video games. By using occupational activities, participants did weight shifting in the sagittal and frontal planes. The investigators also used a balance board (Reebok Core board) for multi-directional weight shifting training
  Interventions: Other: Conventional weight-shifting(30 Mins)

INTERVENTIONS:
Device: Wii Fit(30 Mins) — Receive Wi Fit games training for 30 minutes. There are 2 sections for 1 week; the intervention period will be 12 weeks.
  Arms: Wii Fit
Device: Tetrax biofeedback(30 Mins) — Receive Tetrax biofeedback games training for 30 minutes. There are 2 sections for 1 week; the intervention period will be 12 weeks.
  Arms: Tetrax biofeedback
Other: Conventional weight-shifting(30 Mins) — Receive weight-shifting exercise training for 30 minutes. There are 2 sections for 1 week; the intervention period will be 12 weeks.
  Arms: Conventional weight-shifting

SUMMARY:
The objective of this study was to: compare the training and maintenance effects of 3 balance training programs (2 kinds of exergame systems and 1 conventional weight-shifting training program) on cognitive function of subjects with chronic stroke.

DETAILED DESCRIPTION:
The objective of this study was to: compare the training and maintenance effects of 3 balance training programs (2 kinds of exergame systems and 1 conventional weight-shifting training program) on cognitive function of subjects with chronic stroke. We hypothesized that the exergaming program using weight shifting as game controller is better than the weight shifting only program. The investigators further hypothesized that exergames designed for entertainment (such as Wii Fit) are more beneficial than exergames for rehabilitation purpose (such as Tetrax biofeedback) in gain of cognition function for patients with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Post-stroke duration of at least 6 months
* Ability to understand verbal instructions and learn
* Adequate visual acuity (with appropriate correction, if necessary)
* Ability to walk independently with or without device

Exclusion Criteria:

* Bilateral hemispheric
* Cerebellar lesions
* Aphasia
* Significant visual field deficits
* Hemineglect
* History of orthopedic
* Other neurological diseases
* Medical conditions that would prevent adherence to the exercise protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Cognitive Abilities Screening Instrument Scale Chinese version (CASI C-2.0) | Subjects will be assesed at 12 weeks and 24 weeks
  The CASI C-2.0 consists of 20 item sets, which can be divided into 9 domains, including long-term memory, short-term memory, attention, concentration or mental manipulation, orientation, abstraction/judgment, language, visual construction, and category fluency. The CASI scores range from 0 to 100, with higher scores indicating better cognitive performance.

SECONDARY OUTCOMES:
Change from Baseline in The Stroop test | Subjects will be assesed at 12 weeks and 24 weeks
  The Stroop test requires selective attention, response inhibition, and working memory. The Stroop score ranges from 0 to 63, with higher scores indicating better performance.
Change from Baseline in The modified Trail Making Test(TMT) | Subjects will be assesed at 12 weeks and 24 weeks
  The modified Trail Making Test (TMT) requires visual scanning, visuo-motor tracking, divided attention, and cognitive flexibility. The shorter time to complete the test means better performance.
Change from Baseline in The digit backward performance | Subjects will be assesed at 12 weeks and 24 weeks
  The digit backward performance requires attention and working memory. The scores range from 2 to 7 higher scores indicating better performance.
Change from Baseline in Physiological profile assessment(PPA) | Subjects will be assesed at 12 weeks and 24 weeks
  The PPA is a validated battery of sensorimotor measurements used to identify those subjects at risk of falling.
Change from Baseline in The 10m walking test | Subjects will be assesed at 12 weeks and 24 weeks
  The 10m WT is a reliable, valid, and responsive measure for sub-acute stroke. Walking speed will be assessed by self-selected gait speed over 10 m. The shorter time it takes is indicating better performance.
Change from Baseline in Tetrax balance system | Subjects will be assesed at 12 weeks and 24 weeks
  Tetrax balance system will be used to assess static standing balance. The lower risk scores is indicating better performance.
Change from Baseline in Timed Up and Go (TUG) test | Subjects will be assesed at 12 weeks and 24 weeks
  Timed Up and Go (TUG) test will be used to assessed Dynamic balance function. The shorter time it take means better performance.
Change from Baseline in The Frenchay Activities Index (FAI) | Subjects will be assesed at 12 weeks and 24 weeks
  The Frenchay Activities Index (FAI) was used as a measure of subjects' participation level. The 15-item index records the frequency of performing social activities as well as more complex activities of daily living (eg, domestic chores, outdoor mobility, leisure, gainful work). The FAI item score is based on the frequency with which an activity was performed, and ranges from 0 (low frequency) to 3 (high frequency). Ten items concern the past 3 months and 5 items concern the past 6 months. The FAI total score is the sum of item scores, and ranges from 0 (inactive) to 45 (highly active).
Change from Baseline in Stroke Impact Scale | Subjects will be assesed at 12 weeks and 24 weeks
  The Stroke Impact Scale (SIS) is a 59-item self-reported scale with good reliability, validity, and sensitivity to change. The SIS consists of 8 functional domains: strength, memory, emotion, communication, ADL/ instrumental ADL (IADL), mobility, hand function, and participation. The overall SIS score represents the average score of the 8 domains. Each item score ranges from 1 to 5. Each domain score has a range of 0 to 100 and is computed by using the following equation: Score =[(Mean - 1)/(5 - 1)] × 100. In this equation, the score is that of a particular domain, and the mean is the average of the item scores within that domain. A higher score on an item denotes better performance.
Change from Baseline in Physical Activity Enjoyment Scale (PACES) | Subjects will be assesed at 12 weeks and 24 weeks
  The PACES is a 18-item and 7-point self-reported scale, and the higher score has more enjoyment of the training.

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Wen Hung, MD, Principal Investigator — Chang Gung Memorial Hospital-Kaohsiung Medical Center, Kaohsiung, Taiwan
Locations (1):
- Department of Rehabilitation, Chang Gung Memorial Hospital-Kaohsiung Medical Center, Kaohsiung, Taiwan, Kaohsiung, Taiwan, Taiwan

REFERENCES:
- [Background] Zinn S, Dudley TK, Bosworth HB, Hoenig HM, Duncan PW, Horner RD. The effect of poststroke cognitive impairment on rehabilitation process and functional outcome. Arch Phys Med Rehabil. 2004 Jul;85(7):1084-90. doi: 10.1016/j.apmr.2003.10.022. PMID 15241754
- [Background] Mok VC, Wong A, Lam WW, Fan YH, Tang WK, Kwok T, Hui AC, Wong KS. Cognitive impairment and functional outcome after stroke associated with small vessel disease. J Neurol Neurosurg Psychiatry. 2004 Apr;75(4):560-6. doi: 10.1136/jnnp.2003.015107. PMID 15026497
- [Background] Nys GM, van Zandvoort MJ, de Kort PL, Jansen BP, de Haan EH, Kappelle LJ. Cognitive disorders in acute stroke: prevalence and clinical determinants. Cerebrovasc Dis. 2007;23(5-6):408-16. doi: 10.1159/000101464. Epub 2007 Apr 2. PMID 17406110
- [Background] Nys GM, van Zandvoort MJ, de Kort PL, van der Worp HB, Jansen BP, Algra A, de Haan EH, Kappelle LJ. The prognostic value of domain-specific cognitive abilities in acute first-ever stroke. Neurology. 2005 Mar 8;64(5):821-7. doi: 10.1212/01.WNL.0000152984.28420.5A. PMID 15753416
- [Background] Tatemichi TK, Paik M, Bagiella E, Desmond DW, Pirro M, Hanzawa LK. Dementia after stroke is a predictor of long-term survival. Stroke. 1994 Oct;25(10):1915-9. doi: 10.1161/01.str.25.10.1915. PMID 8091433
- [Background] Hobson P, Meara J. Cognitive function and mortality in a community-based elderly cohort of first-ever stroke survivors and control subjects. J Stroke Cerebrovasc Dis. 2010 Sep-Oct;19(5):382-7. doi: 10.1016/j.jstrokecerebrovasdis.2009.07.006. Epub 2010 May 15. PMID 20472471
- [Background] Pasquini M, Leys D, Rousseaux M, Pasquier F, Henon H. Influence of cognitive impairment on the institutionalisation rate 3 years after a stroke. J Neurol Neurosurg Psychiatry. 2007 Jan;78(1):56-9. doi: 10.1136/jnnp.2006.102533. Epub 2006 Sep 4. PMID 16952914
- [Background] Pollock A, St George B, Fenton M, Firkins L. Top ten research priorities relating to life after stroke. Lancet Neurol. 2012 Mar;11(3):209. doi: 10.1016/S1474-4422(12)70029-7. No abstract available. PMID 22341029
- [Background] Rand D, Eng JJ, Liu-Ambrose T, Tawashy AE. Feasibility of a 6-month exercise and recreation program to improve executive functioning and memory in individuals with chronic stroke. Neurorehabil Neural Repair. 2010 Oct;24(8):722-9. doi: 10.1177/1545968310368684. Epub 2010 May 11. PMID 20460494
- [Background] Quaney BM, Boyd LA, McDowd JM, Zahner LH, He J, Mayo MS, Macko RF. Aerobic exercise improves cognition and motor function poststroke. Neurorehabil Neural Repair. 2009 Nov;23(9):879-85. doi: 10.1177/1545968309338193. Epub 2009 Jun 18. PMID 19541916
- [Background] Marzolini S, Oh P, McIlroy W, Brooks D. The effects of an aerobic and resistance exercise training program on cognition following stroke. Neurorehabil Neural Repair. 2013 Jun;27(5):392-402. doi: 10.1177/1545968312465192. Epub 2012 Nov 16. PMID 23161865
- [Background] Feng J, Spence I, Pratt J. Playing an action video game reduces gender differences in spatial cognition. Psychol Sci. 2007 Oct;18(10):850-5. doi: 10.1111/j.1467-9280.2007.01990.x. PMID 17894600
- [Background] Green CS, Bavelier D. Action video game modifies visual selective attention. Nature. 2003 May 29;423(6939):534-7. doi: 10.1038/nature01647. PMID 12774121
- [Background] Franceschini S, Gori S, Ruffino M, Viola S, Molteni M, Facoetti A. Action video games make dyslexic children read better. Curr Biol. 2013 Mar 18;23(6):462-6. doi: 10.1016/j.cub.2013.01.044. Epub 2013 Feb 28. PMID 23453956
- [Background] Lieberman DA. Designing serious games for learning and health in informal and formal settings. In: Ritterfeld U, Cody MJ, Vorderer P, editors. Serious games: mechanisms and effects. New York: Routledge; 2009. p 117-30.
- [Background] O'Leary KC, Pontifex MB, Scudder MR, Brown ML, Hillman CH. The effects of single bouts of aerobic exercise, exergaming, and videogame play on cognitive control. Clin Neurophysiol. 2011 Aug;122(8):1518-25. doi: 10.1016/j.clinph.2011.01.049. Epub 2011 Feb 24. PMID 21353635
- [Background] Padala KP, Padala PR, Malloy TR, Geske JA, Dubbert PM, Dennis RA, Garner KK, Bopp MM, Burke WJ, Sullivan DH. Wii-fit for improving gait and balance in an assisted living facility: a pilot study. J Aging Res. 2012;2012:597573. doi: 10.1155/2012/597573. Epub 2012 Jun 13. PMID 22745909
- [Background] Rosenberg D, Depp CA, Vahia IV, Reichstadt J, Palmer BW, Kerr J, Norman G, Jeste DV. Exergames for subsyndromal depression in older adults: a pilot study of a novel intervention. Am J Geriatr Psychiatry. 2010 Mar;18(3):221-6. doi: 10.1097/JGP.0b013e3181c534b5. PMID 20173423
- [Background] Zimmermann R, Gschwandtner U, Benz N, Hatz F, Schindler C, Taub E, Fuhr P. Cognitive training in Parkinson disease: cognition-specific vs nonspecific computer training. Neurology. 2014 Apr 8;82(14):1219-26. doi: 10.1212/WNL.0000000000000287. Epub 2014 Mar 12. PMID 24623840
- [Background] Lohse K, Shirzad N, Verster A, Hodges N, Van der Loos HF. Video games and rehabilitation: using design principles to enhance engagement in physical therapy. J Neurol Phys Ther. 2013 Dec;37(4):166-75. doi: 10.1097/NPT.0000000000000017. PMID 24232363
- [Background] Hung JW, Chou CX, Hsieh YW, Wu WC, Yu MY, Chen PC, Chang HF, Ding SE. Randomized comparison trial of balance training by using exergaming and conventional weight-shift therapy in patients with chronic stroke. Arch Phys Med Rehabil. 2014 Sep;95(9):1629-37. doi: 10.1016/j.apmr.2014.04.029. Epub 2014 May 23. PMID 24862764
- [Background] Teng EL, Hasegawa K, Homma A, Imai Y, Larson E, Graves A, Sugimoto K, Yamaguchi T, Sasaki H, Chiu D, et al. The Cognitive Abilities Screening Instrument (CASI): a practical test for cross-cultural epidemiological studies of dementia. Int Psychogeriatr. 1994 Spring;6(1):45-58; discussion 62. doi: 10.1017/s1041610294001602. PMID 8054493
- [Background] Tsai RC, Lin KN, Wang HJ, Liu HC. Evaluating the uses of the total score and the domain scores in the Cognitive Abilities Screening Instrument, Chinese version (CASI C-2.0): results of confirmatory factor analysis. Int Psychogeriatr. 2007 Dec;19(6):1051-63. doi: 10.1017/S1041610207005327. Epub 2007 Apr 23. PMID 17451615
- [Background] Cumming TB, Tyedin K, Churilov L, Morris ME, Bernhardt J. The effect of physical activity on cognitive function after stroke: a systematic review. Int Psychogeriatr. 2012 Apr;24(4):557-67. doi: 10.1017/S1041610211001980. Epub 2011 Oct 14. PMID 21996131
- [Background] Hung JW, Liou CW, Wang PW, Yeh SH, Lin LW, Lo SK, Tsai FM. Effect of 12-week tai chi chuan exercise on peripheral nerve modulation in patients with type 2 diabetes mellitus. J Rehabil Med. 2009 Nov;41(11):924-9. doi: 10.2340/16501977-0445. PMID 19841845
- [Background] Wayne PM, Walsh JN, Taylor-Piliae RE, Wells RE, Papp KV, Donovan NJ, Yeh GY. Effect of tai chi on cognitive performance in older adults: systematic review and meta-analysis. J Am Geriatr Soc. 2014 Jan;62(1):25-39. doi: 10.1111/jgs.12611. Epub 2014 Jan 2. PMID 24383523
- [Background] D'Angelo E. Neural circuits of the cerebellum: hypothesis for function. J Integr Neurosci. 2011 Sep;10(3):317-52. doi: 10.1142/S0219635211002762. PMID 21960306
- [Background] Zinn S, Bosworth HB, Hoenig HM, Swartzwelder HS. Executive function deficits in acute stroke. Arch Phys Med Rehabil. 2007 Feb;88(2):173-80. doi: 10.1016/j.apmr.2006.11.015. PMID 17270514
- [Background] Galski T, Bruno RL, Zorowitz R, Walker J. Predicting length of stay, functional outcome, and aftercare in the rehabilitation of stroke patients. The dominant role of higher-order cognition. Stroke. 1993 Dec;24(12):1794-800. doi: 10.1161/01.str.24.12.1794. PMID 8248957
- [Background] Zelinski EM, Reyes R. Cognitive benefits of computer games for older adults. Gerontechnology. 2009 Fall;8(4):220-235. doi: 10.4017/gt.2009.08.04.004.00. PMID 25126043
- [Background] Anderson-Hanley C, Arciero PJ, Brickman AM, Nimon JP, Okuma N, Westen SC, Merz ME, Pence BD, Woods JA, Kramer AF, Zimmerman EA. Exergaming and older adult cognition: a cluster randomized clinical trial. Am J Prev Med. 2012 Feb;42(2):109-19. doi: 10.1016/j.amepre.2011.10.016. PMID 22261206
- [Background] Maillot P, Perrot A, Hartley A. Effects of interactive physical-activity video-game training on physical and cognitive function in older adults. Psychol Aging. 2012 Sep;27(3):589-600. doi: 10.1037/a0026268. Epub 2011 Nov 28. PMID 22122605
- [Background] Yong Joo L, Soon Yin T, Xu D, Thia E, Pei Fen C, Kuah CW, Kong KH. A feasibility study using interactive commercial off-the-shelf computer gaming in upper limb rehabilitation in patients after stroke. J Rehabil Med. 2010 May;42(5):437-41. doi: 10.2340/16501977-0528. PMID 20544153
- [Background] Fabel K, Kempermann G. Physical activity and the regulation of neurogenesis in the adult and aging brain. Neuromolecular Med. 2008;10(2):59-66. doi: 10.1007/s12017-008-8031-4. Epub 2008 Feb 20. PMID 18286387
- [Background] Olson AK, Eadie BD, Ernst C, Christie BR. Environmental enrichment and voluntary exercise massively increase neurogenesis in the adult hippocampus via dissociable pathways. Hippocampus. 2006;16(3):250-60. doi: 10.1002/hipo.20157. PMID 16411242
- [Background] Ballesteros S, Mayas J, Prieto A, Toril P, Pita C, Laura Pde L, Reales JM, Waterworth JA. A randomized controlled trial of brain training with non-action video games in older adults: results of the 3-month follow-up. Front Aging Neurosci. 2015 Apr 14;7:45. doi: 10.3389/fnagi.2015.00045. eCollection 2015. PMID 25926790
- [Background] Bossers WJ, van der Woude LH, Boersma F, Hortobagyi T, Scherder EJ, van Heuvelen MJ. A 9-Week Aerobic and Strength Training Program Improves Cognitive and Motor Function in Patients with Dementia: A Randomized, Controlled Trial. Am J Geriatr Psychiatry. 2015 Nov;23(11):1106-16. doi: 10.1016/j.jagp.2014.12.191. Epub 2015 Jan 3. PMID 25648055
- See also: Nintendo. Nintendo Wii-Fit games — http://www.nintendo.com/